CLINICAL TRIAL: NCT05197478
Title: LIFE STYLE BEFORE COVID 19 INFECTION IMPACT ON THE PROGRESS OF COVID 19
Brief Title: THE EFFECT OF LIFESTYLE ON THE PROGRESS OF COVID 19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: yildizyigit1
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Lifestyle Factors
Keywords: COVİD 19; LİFESTYLE; PANDEMİA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: It was conducted prospectively on 31 January - 31 May 2021 patients over 50 years of age, who were hospitalized in the pandemic ward, had the appearance of COVID 19, and were taken into ethical examination (E-17073117-050.06). 50.06,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID 19 positive patients (Other): COVID 19 positive patients receiving inpatient treatment were evaluated.
  Interventions: Other: Mini Nutritional Assessment ,Pıtsburg Sleep Qualıty Scale, Short Physical Activity Survey

INTERVENTIONS:
Other: Mini Nutritional Assessment ,Pıtsburg Sleep Qualıty Scale, Short Physical Activity Survey — To evaluate the lifestyle before being infected with COVID 19, physical activity, nutrition and sleep habits were questioned.
  To evaluate sleep habits; Pitsburg Sleep Quality Scale (PSQS) Nutritional habits: Mini Nutritional Assessment(MNA) Scale For the evaluation of physical activity; International Brief Physical Activity Questionnaire

SUMMARY:
THE EFFECT OF LIFESTYLE ON THE PROGRESS OF COVID 19 INFECTION

The development of COVID 19 disease depends on the interaction with the immunity of the host. The immune response of the host is related to age, gender, nutrition, sleep and physical activity. Our study in Fatih Sultan Mehmet Training and Research Hospital; Between 31 January-31 May 2021,positive COVID 19 PCR test was performed with 66 patients over the age of 50, who received inpatient treatment. Demographic data of the patients, length of hospitalization, alcohol/tobacco use, BMI, comorbidities, regular use medication or not, thorax CT findings, place of discharge after treatment, laboratory parameters were recorded at hospitalization and discharge.

To evaluate the pre-infection lifestyle; physical activity, nutrition and sleep habits were questioned.

According to the PSQS (Pittsburg Sleep Quality Scale) although the increase in discharged lymphocyte measurements compared to the first hospitalization of the patients in the good and bad sleep groups was significant, there was no significant difference between the groups. In the evaluation between the groups, the increase in the NLR value at the first hospitalization was significant in the bad sleep group compared to the good sleep group. There was no difference between the groups in terms of NLR.

According to the MNA(Mini Nutritional Assessment)scale ;the increase in the discharge lymphocyte value of the groups compared to the value at the first hospitalization was significant. The increases in the discharge lymphocyte measurements of the patients compared to the first hospitalization were significant between the groups (p<0.05). The increase in discharge lymphocyte values in patients at risk of malnutrition compared to the first hospitalization was higher than in patients with malnutrition (p<0.05). The decrease in discharge NLR values compared to the first hospitalization was significant in the group under normal nutrition and malnutrition risk. The difference between the first hospitalization PLT (Platelet)measurements of the groups according to the MNA scale was significant.

According to the International Brief Physical Activity Survey; the increase in the discharge lymphocyte value of the inactive, minimally active and very active groups was significant compared to the first hospitalization. A significant difference was found between the PLT measurements between the groups (p<0.05). PLT measurements of very active cases were higher than those of minimally active cases (p<0.05).

In this study, in which we examined the effects of lifestyle before the diagnosis of COVID 19 on the course of COVID 19, we observed that there is no need for intensive care in patients who are well fed, have good sleep quality and are physically active.

DETAILED DESCRIPTION:
Our study in Fatih Sultan Mehmet Training and Research Hospital; It was conducted prospectively on 31 January - 31 May 2021:

Inclusion criteria:

Patients over 50 years of age, Who were hospitalized in the pandemic ward Patients with positive COVID 19 pcr test and were taken into ethical examination (E-17073117-050.06)

Exclusion criteria:

Patients under 50 years of age, Patients with negative COVID 19 pcr test, Lymphatic system disease or malignant hematological diseases were excluded from the study.

Patient age, gender, education status,time spent at home before hospitalization ,duration of hospitalization, alcohol/tobacco use, body mass index,presence of thorax CT lesion ,whether the patients were discharged to another service, intensive care unit, or home after the treatment of COVID 19,laboratory findings at admission and discharge (lymphocyte level, neutrophil-lymphocyte ratio and platelet count at first admission) were recorded.

To evaluate the lifestyle before being infected with COVID 19, physical activity, nutrition and sleep habits were questioned.

To evaluate sleep habits; Pittsburg Sleep Quality Scale (PSQS) , Nutritional habits; Mini Nutritional Assessment(MNA) Scale, For the evaluation of physical activity; International Brief Physical Activity Questionnaire Done.

ELIGIBILITY:
Inclusion Criteria:

COVID 19 pcr test positive over 50 years of age, inpatient treatment patients with pandemic service received ethics committee approval

Exclusion Criteria:

COVID 19 pcr negative Under 50 years of age, Lymphatic system patients with disease or malignant hematological diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) . | UP TO 24 WEEKS
  SLEEP QUALİTY SCALE The total PSQI score is obtained by summing the seven sub-scores. The total score ranges from 9 to 21. The PSQI total score clearly distinguishes good sleepers from bad sleepers.
  Good sleep:5 points or less Bad Sleep:over 5 points
Mini Nutritional Assessment | UP TO 24 WEEKS
  NUTRITIONAL STATUS
  The sum of the MNA score distinguishes between elderly patients with:
  1. Adequate nutritional status, MNA 24;
  2. Protein-calorie malnutrition, MNA 17;
  3. at risk of malnutrition, MNA between 17 and 23.5.
  Normal nutritional status:24-30 points
  At risk of malnutrition:17-23.5
  Malnourished:under 17 points
International Short Physical Activıiy Questionnaire | UP TO 24 WEEKS
  Category 1:INACTIVE
  It is the lowest level of physical activity. Conditions that cannot be included in categories 2 and 3 are considered inactive.
  Category 2:MINIMUM ACTIVE
  2 a:Doing vigorous activity for at least 20 minutes on 3 or more days 2b:5 or more days of moderate-intensity activity or walking for at least 30 minutes a day
  2c:A combination of 5 or more days of walking and moderate-intensity activity providing a minimum of 600 MET-min/week
  Category 3:VERY ACTIVE
  3 a:At least 3 days of vigorous physical activity or more days providing a minimum of 1500 MET-min/week
  3b:Moderate to vigorous walking for 7 days providing a minimum of 3000 MET-min/week combination of activity

SECONDARY OUTCOMES:
LYMPHOCYTE COUNT | UP TO 24 WEEKS
  HEMATOLOGICAL BIOMARKER
NEUTROPHIL LYMPHOCYTE RATIO | UP TO 24 WEEKS
  HEMATOLOGICAL BIOMARKER
PLATELET COUNT | UP TO 24 WEEKS
  HEMATOLOGICAL BIOMARKER

CONTACTS AND LOCATIONS:
Locations (1):
- Yıldız, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared if requested by the editor.